CLINICAL TRIAL: NCT07197723
Title: Effect of Polygenic Risk Modifiers on Decisions of BRCA1/2 Mutation Carriers at Risk for Prostate Cancer
Brief Title: Study of How People Make Decisions About Prostate Cancer Risk
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: CureBRCA Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 25-235
Record Dates: First submitted 2025-09-25; First posted 2025-09-29 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: BRCA1/2; Geneitic Testing
Keywords: Polygenic Risk Modifiers; BRCA1/2 Mutation Carriers; Assessments

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cheek (buccal) swab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men with BRCA1/2 mutations who are at risk for prostate cancer: Will be offered genetic risk modifier testing (note that this testing is of clinical grade but is not yet standard of care and is therefore only available through the context of this research study), and will complete baseline and then 1-week, 6-month, and 12-month post-receipt of modifier results follow-up quantitative assessments of their psychological and behavioral outcomes.
  Interventions: Genetic: cheek (buccal) swab; Other: Assessments; Other: optional collection of blood

INTERVENTIONS:
Genetic: cheek (buccal) swab — swab sample in person or at home with a mailed test kit and will fill out a survey
Other: Assessments — about 1 week, 6 months, and 12 months after getting the updated cancer risk assessment to complete additional surveys.
Other: optional collection of blood — for research testing

SUMMARY:
The purpose of this study is to learn how people with BRCA1/2 mutations respond to genetic risk modifier testing. The researchers will learn more about how people make choices about their health care, including about methods to screen for prostate cancer. Researchers are also doing this study to learn about how the genetic risk modifier test affects people's thoughts and feelings.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of Disease

  o Patients must not have prostate cancer
* Age between 45 - 70;
* Assigned male sex at birth
* Completed full sequence or targeted genetic testing with a result confirmed in a clinically approved laboratory showing a BRCA1/2 likely pathogenic or pathogenic variant identified
* English-fluent; the surveys were designed and validated in English and are not currently available in other languages. Translation of questionnaires into other languages would require reestablishing the reliability and validity of these measures. Therefore, participants must be able to communicate in English to complete the surveys.

Exclusion Criteria:

* Major psychiatric illness or cognitive impairment that in the judgment of the study investigators or study staff would preclude study participation.
* Any patients who are unable to comply with the study procedures as determined by the study investigators or study staff.
* Under active treatment for a malignancy. (Patients are eligible if they have a prior history of malignancy other than prostate cancer, as long as they are not currently undergoing active treatment for the malignancy)
* Enrolled in NCI study 19-C-0040 (Natural History of Men at High-Risk for Prostate Cancer) based on self-report

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Study Population: Potential participants (i.e., male MSK patients with a documented BRCA1/2 PV) will be identified by study staff who will screen relevant clinic schedules (e.g., for the MSK CATCH high-risk screening clinic, for post-test visits in the MSK CGS) and approached by their clinician (primary genetic counselor, and/or clinician in the high-risk screening clinic or other MSK clinician) with support from study staff.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Intention to undergo prostate cancer screening options | 6 months
  Change in intention for each screening option measured with the Choice predisposition scale. Choice Predisposition scale ranges from 1 (leaning towards yes) to 15 (leaning towards no) regarding a specific option.

CONTACTS AND LOCATIONS:
Overall Officials: Jada Hamilton, PhD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm